CLINICAL TRIAL: NCT06440733
Title: Effectiveness of 8 Week Multicomponent Exercise Program on the General Health and Balance of a Group of Older Adults With Frailty and Cognitive Impairment: a Quasi-experimental Pilot Study
Brief Title: Effectiveness of 8 Week Multicomponent Exercise Program in Older Adults With Frailty and Cognitive Impairment
Acronym: GERYPHYSIO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Rocío Martín Valero, Principal Investigator, University of Malaga
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMalagaGER
Record Dates: First submitted 2024-05-23; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Old Age; Debility
Keywords: Multicomponent exercise program; Fragility; Elderly; Balance; Quality of life; Autonomy; Functionality
MeSH Terms: conditions — Frailty | interventions — Aging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Older adults with frailty and cognitive impairment (Experimental): In this study, an 8-week multicomponent exercise program will be carried out focused on improving the general physical condition and balance of older adult subjects, in order to try to reduce the risk of falls and improve the quality of life of a group. of older adults made up of 17 participants.
  Interventions: Other: Multicomponent exercise program focused in elderly.

INTERVENTIONS:
Other: Multicomponent exercise program focused in elderly. — Each of these sessions will be carried out taking into account the main physiotherapy objectives, such as gaining strength in both upper and lower limbs, as well as proprioception, balance, and promoting a pleasant and safe social environment where these older people feel valid.
  All sessions will begin with a 5-minutes. It will begin with a general warm-up based on general joint mobility of the head and neck, shoulders, trunk, elbows, hands, wrists, hips, knees and ankles to begin to accustom the body to the physical work environment. And at the end of the sessions, a stretching program will be carried out, and it will end with a return to calm with a respiratory training program, in which you will be instructed to take in air through the nose and release it through the mouth, while the room is silent, and thus promote self-awareness.

SUMMARY:
Multicomponent exercise program in a frail population. It is analyzed whether there is an improvement in different parameters of the daily life of the study subjects, analyzing the variables of: physical condition, fragility, balance, quality of life, upper limb strength, autonomy, cognitive state and depression.

DETAILED DESCRIPTION:
In this study, an 8-week multicomponent exercise program will be carried out focused on improving the general physical condition and balance of older adult subjects, in order to try to reduce the risk of falls and improve the quality of life of a group. of older adults made up of 17 participants.

During these 8 weeks, this intervention program will be carried out at least 3 times a week, for 50-55 minutes, which will consist of 4 typical sessions, based mainly on 5 large groups: weights, magic rings, elastic bands, ballasts and pikes... Each of these sessions will be carried out taking into account the main physiotherapy objectives, such as gaining strength in both upper and lower limbs, as well as proprioception, balance, and promoting a pleasant and safe social environment where these older people feel valid, capable of carrying out the program and everything is provided to them in a friendly and fun way, and always taking into account as far as possible , the individual characteristics of each study participant. All sessions will begin with a 5-minute aerobic exercise and end with a stretching program for another 5 minutes, to ensure you return to calm, along with breathing exercises.

The intervention will begin by carrying out an initial evaluation already developed previously, and after this, standard sessions will begin, in which they will all begin and end in the same way. It will begin with a general warm-up based on general joint mobility of the head and neck, shoulders, trunk, elbows, hands, wrists, hips, knees and ankles to begin to accustom the body to the physical work environment. And at the end of the sessions, a stretching program will be carried out, and it will end with a return to calm with a respiratory training program, in which you will be instructed to take in air through the nose and release it through the mouth, while the room is silent, and thus promote self-awareness.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 65 years of age.
* People with frailty according to the Short Physical Performance Battery,
* who have the ability to walk (autonomous or with external aids),
* and who obtain a score greater than or equal to 15 in the Lobo Mini Cognitive Examination (MEC-35 of Lobo).
* patients with a resolved hip fracture, with Parkinson's,
* Patients who are committed and motivated to carry out the study, as well as patients who agree to sign the informed consent and the report sheet prior to carrying out the study.

Exclusion Criteria:

* Old Adults under 65 years of age.
* Patients who do not present frailty or the ability to walk (autonomous or with external aids).
* People who obtain a score of less than 15 in the Lobo Mini Cognitive Exam therefore presenting a serious deterioration of the emotional and cognitive state.
* Older adults who are under treatment with tranquilizers or sedatives, non-diuretic hypotensive agents or antidepressants.
* Patients with amyotrophic lateral sclerosis, multiple sclerosis, diabetic neuropathy, severe sensory deficit, and study subjects without motivation or interest in participating in the study.
* Older adults who do not agree to sign the study, will also be excluded from the study. informed consent and the report sheet prior to carrying out the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2023-09-30 (Actual); Primary Completion 2024-08-19 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Short Physical Performance Battery | Baseline up to 8 weeks.
  Analyze if there are changes in general physical condition and frailty after an 8 week multicomponent exercise program in a group of older adults before and after carrying it out using the Short Physical Performance Battery questionnaire. The score obtained with this geriatric evaluation test ranges between 0 and 12 points, and can be interpreted depending on the result obtained as: severe limitation or disabled between 0-3, moderate limitation or fragile/vulnerable between 4-6, limitation mild or pre-frail between 7-9, minimal limitation or autonomous/healthy between 10-12. However, if the participant obtains a score of less than 10 on the SPPB, it can be used as a mortality assessment criterion in studies that need to quantify the health benefits and improvements of specific treatments or rehabilitation programs, such as case of this present study.
Tinetti scale | Baseline up to 8 weeks
  Analyze the risks of falling before performing the multicomponent exercise program and after it, seeing if there is variation in it in the group of older adults using the Tinetti scale for balance and gait. The maximum score achievable with this scale is 28 points and 16 of them coming from the balance sphere, and 12 points coming from the gait sphere. So: High risk of falling: score less than 19 points, Average risk of falling: 19 to 23 points, and Low risk of falling: 24 to 28 points.

SECONDARY OUTCOMES:
Short Form 12 Questionnaire | Baseline, up to 8 weeks.
  Check the influence of the multicomponent exercise program on the quality of life of the group of older adults using the Short-Form questionnaire . In this study, a variant of the questionnaire will be used in which Z scores are provided, that is, scores that compare with the average of the population, in this case comparing with the American population, being in both cases an average of 50. Everything that is close to 50 will be considered standard quality of life, everything that is above 50 will be considered good quality of life and everything that is below 50 will be considered bad quality of life.
Strength in hands. | Baseline, up to 8 weeks.
  Analyze changes in the muscle strength of the upper limbs of a group of older adults before and after the multicomponent exercise program using a Jamar hand-held dynamometer. To analyze the muscular strength of the upper limbs of the study subjects, a Jamar dynamometer requested as study material from the University of Malaga will be used, and it will be carried out in a specific pattern. The patient will be placed in a sitting position, with a 90º flexion of the elbow and with the hand making a grip on the handle of the device.
Barthel Index | Baseline, up to 8 weeks.
  Prove the changes in the autonomy of a group of older adults before and after a multicomponent exercise program thanks to the Barthel index for basic activities of daily living. The Barthel index contains 10 items, including bathing, toileting, dressing, feeding, bladder control, toileting, chair or bed transfers, stair climbing, and ambulation. Its items are scored based on the degree of dependence that the patient presents, with a score that can range from 0 to 100, with 0 being a maximum level of dependence and 100 being a maximum level of independence according to the scale.
Yesavage depression scale | Baseline, up to 8 weeks.
  Check the changes at a cognitive, emotional and social level before and after the multicomponent exercise program using Yesavage Geriatric Depression Scale. This scale is scored from 0 to 15, with a score less than 5 being the range of normality, between 5-9 being the range of mild depression, and a score higher than 10 being indicative of moderate to severe depression, being questions with a dichotomous response to items 1, 5, 7, 11, and 13 are considered indicative of depression.
Lobo Mini Cognitive Examination | Baseline, up to 8 weeks.
  Analyze changes at a cognitive, emotional and social level before and after the multicomponent exercise program using Lobo Mini Cognitive Examination. The Lobo Mini Cognitive Examination (MEC) is a test that analyzes the cognitive deterioration of patients, coming from the adaptation of the original test "Mini-Mental State Examination" (MMSE) created by Folstein , performed by Lobo in 1979 .The initial test Mini-Mental State Examination consists of 30 points, unlike the Mini Cognitive Examination, which presents up to a score of 35, analyzing 6 cognitive abilities, plus five more questions on attention, calculation and language, also presenting a completion time of between 10 and 15 minutes. Cognitive impairment is considered to exist when the score is less than 23 points.

CONTACTS AND LOCATIONS:
Overall Officials: Rocío Martín Valero, Study Director — University of Malaga
Locations (1):
- Cristian Carmona Cantalejo, Estación de Cártama, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No